CLINICAL TRIAL: NCT03963271
Title: Noninvasive Electrocardiographic Imaging for Individuals at Risk for Apparently Idiopathic Ventricular Fibrillation.
Acronym: VIGILANCE
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Dutch Heart Foundation (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); UMC Utrecht (Other)
Responsible Party: Sponsor
Other Study IDs: NL67079.068.18
Record Dates: First submitted 2019-04-23; First posted 2019-05-24 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-07

CONDITIONS: Ventricular Fibrillation; Ventricular Arrythmia; Polymorphic Ventricular Tachycardia; Sudden Cardiac Death; Heart Arrest; Cardiovascular Diseases; Cardiac Arrhythmia; Genetic Disease; Idiopathic Ventricular Fibrillation; Cardiac Arrest
Keywords: idiopathic ventricular fibrillation; polymorphic ventricular tachycardia; body surface potential mapping; ECG Imaging
MeSH Terms: conditions — Ventricular Fibrillation; Death, Sudden, Cardiac; Heart Arrest; Cardiovascular Diseases; Arrhythmias, Cardiac; Genetic Diseases, Inborn; Paroxysmal ventricular fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — DNA samples from blood, if analysed upon clinical indication
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with unexplained polymorphic VT and/or VF: 1. Unexplained polymorphic VT and/or VF patients.
  2. Patients with VF and the DPP6 risk haplotype, reported by the AUMC team.
  3. The Worm population of patients with a SCN5A founder mutation and other conspiring genetic variants at MUMC+
  Interventions: Diagnostic Test: ECG-Imaging
- Family members: Family members of index patients of group(s) mentioned above
  Interventions: Diagnostic Test: ECG-Imaging
- Control group: Control subjects with structurally normal hearts with an indication for a cardiac CT,
  Interventions: Diagnostic Test: ECG-Imaging

INTERVENTIONS:
Diagnostic Test: ECG-Imaging — A body surface potential mapping and a cardiac + low dose CT-scan.

SUMMARY:
This study aims to evaluate the electrophysiological properties of the heart conduction system in patients with unexplained polymorphic ventricular tachycardia (VT) and/or ventricular fibrillation (VF), in patients with specific genetic mutations regarding sudden cardiac death or sudden cardiac arrest, in their family members and in a control cohort. The electrophysiological properties will be measured with the relatively new technique ECG-Imaging (ECGI).

Also a National Dutch registry for patients with unexplained polymorphic VT and/or VF and their family members will be created.

By combining the data from the registry and the results of ECGI, The investigators hope to identity risk markers for patients at higher risk for apparently idiopathic ventricular fibrillation, and use these for an adapted flow chart for the 'general'population of patients at risk for unexplained polymorphic VT and/or VF. The investigators aim to be able to identify patients before the first arrhythmic event, and aim for better treatment strategies in the future.

DETAILED DESCRIPTION:
ECGI combines electrical body-surface mapping with 256 electrodes placed on the thorax with a CT-scan obtaining the anatomy of the heart and torso, hereby able to reconstruct local electrograms, activation and recovery times. In recent research, ECGI provided numerous extra insights into normal cardiac electrophysiology, but also electrophysiological disorders and disease. The results strongly suggest that ECGI can play a pivotal role in further characterizing arrhythmia mechanisms, therefore could do so for polymorphic VT or idiopathic VF leading to diagnosis and treatment improvement. Moreover, ECGI seems to have the potential to detect arrhythmogenic substrate in individuals before their first event, offering the possibility to diagnose and treat patients before sudden cardiac arrest occurs.

In the VIGILANCE study:

1. ECGI will be used to noninvasively characterize the epicardial electrophysiological substrate and triggers of:

   * Patients with unexplained polymorphic VT and VF,
   * Index patients of family cohorts with a specific genetic mutation related to arrhythmogenesis, at high risk for unexplained polymorphic VT and/or VF.
   * Family members,
   * A control cohort. Results will be evaluated for risk stratification.
2. All unexplained polymorphic VT and/or VF patients and their family members will be asked to participate in a National Dutch registry, and these date will be analysed to determine their prognostic value in terms of arrhythmia risk

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, a subject must be ≥ 18 years old and meet one of the following criteria:

* All unexplained polymorphic VT or VF survivors in whom known structural myocardial, respiratory, metabolic and toxicological causes have been excluded through clinical evaluation", with/without a genetic mutation. NB. If results of a diagnostic tests show minor abnormalities but insufficient for a specific diagnosis, this is no exclusion criterion.
* Selected family members of these patients*
* Control subjects with structurally normal hearts with a clinical indication for a cardiac CT scan.

  * All 1st and 2nd degree family members being in contact with the cardiologist/treating physician as part of cascade screening will be contacted as described in chapter 11.2.2.

Family members must be in adequate health to be able to travel to the hospital for research purposes.

3rd degree family members can also be contacted as described in chapter 11.2.2 if at least one of the following criteria is met:

* The family member has the same genetic mutation as index patient, or;
* The family member has demonstrated ventricular arrhythmias, or;
* The clinician has a very strong suspicion of ventricular arrhythmias in the family member.

Exclusion Criteria:

A potential subject who meets any of the following criteria will be excluded from participation in this study:

* A known strong reaction against electrode attachment or contrast agent.
* Any serious medical condition, which in the opinion of the investigator, may adversely affect the safety and/or effectiveness of the participant or the study.
* Pregnancy, nursing or planning to be pregnant.
* Subject has an estimated glomerular filtration rate (eGFR) of <30mL/min/1.73m2

  , using the MDRD calculation
* Unability to give informed consent.
* Family members of patients with unexplained polymorphic VT/VF, who have severe cardiac abnormalities and/or disease not related to the symptoms or phenotype of the index patient, and which may have a negative influence on results of ECGI according to local investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients seen at the outpatient clinic at the department of cardiology or (cardio)genetics, patients admitted to the ward of cardiology or the intensive care unit.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-04-10 (Actual); Primary Completion 2023-04-10 (Estimated); Study Completion 2023-04-10 (Estimated)

PRIMARY OUTCOMES:
ECG-Imaging outcome: epicardial potentials | 3 years
  reconstructed epicardial potentials, represented in mV over time(s).
ECG-Imaging outcome: activation and repolarization maps | 3 years
  Activation and repolarization maps. These are made by measuring acivation and repolarization times from the reconstructed potentials in miliseconds. Then local activation and recovery times are plotted on a CT-derived heart mesh. The entire activation and repolarization of the epicardium of the heart can be visualized this way.

SECONDARY OUTCOMES:
(Possible) Prognostic risk factors for recurrent ventricular arrhythmias | 3 years
  possible risk factors, found in the registry, given as odds/hazard ratio.
Recurrence of ventricular arrhythmias | 3 years
  documentation over the period of follow-up, if studysubjects had a recurrence of ventricular arrythmia(s), presented as number of events over a time period.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Volders, MD, PhD, Principal Investigator — Maastricht University Medical Centre
Locations (3):
- Netherlands (3):
  - Maastricht Universite Medical Centre, Maastricht, Nederland
  - Amsterdam University medical Centre, location AMC, Amsterdam
  - University Medical Centre Utrecht, Utrecht